CLINICAL TRIAL: NCT01524757
Title: Proton Pump Inhibitors in the Prevention of Iron Reaccumulation in Patient With Hereditary Hemochromatosis
Acronym: He-ppi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Annadal stichting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL3364409612
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Hemochromatosis
MeSH Terms: conditions — Hemochromatosis | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pantoprazol (Experimental)
  Interventions: Drug: Pantoprazole
- placebo (Placebo Comparator)
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — pantoprazole 40mg 1dd1; 12 months

SUMMARY:
Hereditary Hemochromatosis (HH) is a genetic disorder of iron metabolism, resulting in excessive iron overload causing damage of different important organs like heart, liver, pancreas and joints. Complications and symptoms can regress by intensive treatment reducing the iron overload stores.Different genes have been identified playing a role in the pathophysiology of iron overload. A clinically important HFE gene mutation is the C282Y, located on chromosome 6. Phlebotomy is currently the standard therapy which consists of removal of 500 ml whole blood weekly, representing a loss of 250 mg iron. In naive patients between 20 to 100 phlebotomies are required to reduce the serum ferritine levels to 50 μg/L. Thereafter, a lifelong maintenance therapy of 3 to 6 phlebotomies yearly is needed.

For absorption, dietary iron ( 70%) is reduced by gastric acid form the ferric (Fe3+) to the ferrous form (Fe2+). Recently, in an observational open study, Hutchinson et al. found that HH patients treated with proton pump inhibitors (PPI) needed fewer phlebotomies, resulting in a drop of 2.5 (SEM 0.25) to 0.5 (SEM 0.25) liter per year.

Research question: The primary objective is to determine the effectiveness and cost effectiveness of PPI's compared to standard phlebotomy therapy in the prevention of iron overload in HH patients.

Multi-center trial in two hospitals in the South of Limburg (Atrium medical Center, Maastricht university medical center ) and hospital in Belgium (University Hospital Gasthuisberg). The study will be conducted in randomised double blind manner. The follow up will be one year.

Patients are randomized either for the group receiving a PPI or a placebo. Every 2 month the ferritin level is measured and decided if the patient need a phlebotomy (Ferritin >100 µg/L).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hereditary hemochromatosis (HH), homozygous for C282Y, currently treated with phlebotomy as maintenance therapy for at least 12 months with ≥ 3 phlebotomies per year.
* Ferritin level between 50-100 μg/L at start of the inclusion.
* Age: 18 years- 60 years and weight > 50 kg.

Exclusion Criteria:

* Patients receiving other therapies such as chelating therapy or forced dietary regimen.
* Patients younger than 18 years.
* HH patients with excessive overweight (BMI > 35).
* Patients who are mentally incapacitated.
* Women being pregnant or expecting/ planning to become pregnant during the one year period of the study.
* Patients with a malignancy.
* Patients already on PPI treatment.
* Patients who experienced side effects of PPI's.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
the total number of phlebotomies for the group taking PPI treatment compared to the group taking placebo will be the primary endpoint of the study. | 12 months

SECONDARY OUTCOMES:
number of participants with side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: G Koek, Dr, Principal Investigator — Maastricht University Medical Center
Locations (3):
- University hospital Gasthuisberg, Leuven, Limburg, Belgium
- Netherlands (2):
  - Atrium MC Parkstad, Heerlen, Limburg
  - Maastricht university medical center, Maastricht, Limburg

REFERENCES:
- [Background] Hutchinson C, Geissler CA, Powell JJ, Bomford A. Proton pump inhibitors suppress absorption of dietary non-haem iron in hereditary haemochromatosis. Gut. 2007 Sep;56(9):1291-5. doi: 10.1136/gut.2006.108613. Epub 2007 Mar 7. PMID 17344278
- [Background] Adams P, Brissot P, Powell LW. EASL International Consensus Conference on Haemochromatosis. J Hepatol. 2000 Sep;33(3):485-504. doi: 10.1016/s0168-8278(01)80874-6. No abstract available. PMID 11020008
- [Background] Pietrangelo A. Hereditary hemochromatosis. Biochim Biophys Acta. 2006 Jul;1763(7):700-10. doi: 10.1016/j.bbamcr.2006.05.013. Epub 2006 May 27. PMID 16891003
- [Background] van der Plas SM, Hansen BE, de Boer JB, Stijnen T, Passchier J, de Man RA, Schalm SW. Generic and disease-specific health related quality of life of liver patients with various aetiologies: a survey. Qual Life Res. 2007 Apr;16(3):375-88. doi: 10.1007/s11136-006-9131-y. Epub 2006 Nov 25. PMID 17334830
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines for HFE hemochromatosis. J Hepatol. 2010 Jul;53(1):3-22. doi: 10.1016/j.jhep.2010.03.001. Epub 2010 Apr 18. PMID 20471131
- [Background] Jacobs EM, Meulendijks CF, Elving L, van der Wilt GJ, Swinkels DW. Impact of the introduction of a guideline on the targeted detection of hereditary haemochromatosis. Neth J Med. 2005 Jun;63(6):205-14. PMID 16011012
- [Background] Swinkels DW, Janssen MC, Bergmans J, Marx JJ. Hereditary hemochromatosis: genetic complexity and new diagnostic approaches. Clin Chem. 2006 Jun;52(6):950-68. doi: 10.1373/clinchem.2006.068684. Epub 2006 Apr 20. PMID 16627556
- [Background] Rombout-Sestrienkova E, Nieman FH, Essers BA, van Noord PA, Janssen MC, van Deursen CT, Bos LP, Rombout F, van den Braak R, de Leeuw PW, Koek GH. Erythrocytapheresis versus phlebotomy in the initial treatment of HFE hemochromatosis patients: results from a randomized trial. Transfusion. 2012 Mar;52(3):470-7. doi: 10.1111/j.1537-2995.2011.03292.x. Epub 2011 Aug 16. PMID 21848963
- [Background] Hungin AP, Rubin G, O'Flanagan H. Factors influencing compliance in long-term proton pump inhibitor therapy in general practice. Br J Gen Pract. 1999 Jun;49(443):463-4. PMID 10562747
- [Background] Hicken BL, Tucker DC, Barton JC. Patient compliance with phlebotomy therapy for iron overload associated with hemochromatosis. Am J Gastroenterol. 2003 Sep;98(9):2072-7. doi: 10.1111/j.1572-0241.2003.07292.x. PMID 14499790
- [Background] Bonapace ES, Fisher RS, Parkman HP. Does fasting serum gastrin predict gastric acid suppression in patients on proton-pump inhibitors? Dig Dis Sci. 2000 Jan;45(1):34-9. doi: 10.1023/a:1005496907686. PMID 10695611
- [Background] Newman BH. Blood donor complications after whole-blood donation. Curr Opin Hematol. 2004 Sep;11(5):339-45. doi: 10.1097/01.moh.0000142105.21058.96. PMID 15666658
- [Background] HOFSTETTER JR. [Risks in blood-letting in therapy of hemochromatosis]. Gastroenterologia. 1957;87(3-4):186-91. No abstract available. French. PMID 13448264
- [Background] Klinkenberg-Knol EC, Festen HP, Jansen JB, Lamers CB, Nelis F, Snel P, Luckers A, Dekkers CP, Havu N, Meuwissen SG. Long-term treatment with omeprazole for refractory reflux esophagitis: efficacy and safety. Ann Intern Med. 1994 Aug 1;121(3):161-7. doi: 10.7326/0003-4819-121-3-199408010-00001. PMID 8017742
- [Background] Klinkenberg-Knol EC, Nelis F, Dent J, Snel P, Mitchell B, Prichard P, Lloyd D, Havu N, Frame MH, Roman J, Walan A; Long-Term Study Group. Long-term omeprazole treatment in resistant gastroesophageal reflux disease: efficacy, safety, and influence on gastric mucosa. Gastroenterology. 2000 Apr;118(4):661-9. doi: 10.1016/s0016-5085(00)70135-1. PMID 10734017
- [Background] Creutzfeldt W, Lamberts R. Is hypergastrinaemia dangerous to man? Scand J Gastroenterol Suppl. 1991;180:179-91. doi: 10.3109/00365529109093198. PMID 1675024
- [Background] Solcia E, Fiocca R, Havu N, Dalvag A, Carlsson R. Gastric endocrine cells and gastritis in patients receiving long-term omeprazole treatment. Digestion. 1992;51 Suppl 1:82-92. doi: 10.1159/000200921. PMID 1397749
- [Background] Lamberts R, Brunner G, Solcia E. Effects of very long (up to 10 years) proton pump blockade on human gastric mucosa. Digestion. 2001;64(4):205-13. doi: 10.1159/000048863. PMID 11842276
- [Background] Hallerback B, Unge P, Carling L, Edwin B, Glise H, Havu N, Lyrenas E, Lundberg K. Omeprazole or ranitidine in long-term treatment of reflux esophagitis. The Scandinavian Clinics for United Research Group. Gastroenterology. 1994 Nov;107(5):1305-11. doi: 10.1016/0016-5085(94)90531-2. PMID 7926494
- [Background] Lamberts R, Creutzfeldt W, Struber HG, Brunner G, Solcia E. Long-term omeprazole therapy in peptic ulcer disease: gastrin, endocrine cell growth, and gastritis. Gastroenterology. 1993 May;104(5):1356-70. doi: 10.1016/0016-5085(93)90344-c. PMID 8482449
- [Background] Sharma BK, Santana IA, Wood EC, Walt RP, Pereira M, Noone P, Smith PL, Walters CL, Pounder RE. Intragastric bacterial activity and nitrosation before, during, and after treatment with omeprazole. Br Med J (Clin Res Ed). 1984 Sep 22;289(6447):717-9. doi: 10.1136/bmj.289.6447.717. PMID 6434053
- [Background] Fried M, Siegrist H, Frei R, Froehlich F, Duroux P, Thorens J, Blum A, Bille J, Gonvers JJ, Gyr K. Duodenal bacterial overgrowth during treatment in outpatients with omeprazole. Gut. 1994 Jan;35(1):23-6. doi: 10.1136/gut.35.1.23. PMID 8307444
- [Background] Verdu E, Viani F, Armstrong D, Fraser R, Siegrist HH, Pignatelli B, Idstrom JP, Cederberg C, Blum AL, Fried M. Effect of omeprazole on intragastric bacterial counts, nitrates, nitrites, and N-nitroso compounds. Gut. 1994 Apr;35(4):455-60. doi: 10.1136/gut.35.4.455. PMID 8174980
- [Background] Laheij RJ, Sturkenboom MC, Hassing RJ, Dieleman J, Stricker BH, Jansen JB. Risk of community-acquired pneumonia and use of gastric acid-suppressive drugs. JAMA. 2004 Oct 27;292(16):1955-60. doi: 10.1001/jama.292.16.1955. PMID 15507580
- [Background] Koop H, Bachem MG. Serum iron, ferritin, and vitamin B12 during prolonged omeprazole therapy. J Clin Gastroenterol. 1992 Jun;14(4):288-92. doi: 10.1097/00004836-199206000-00005. PMID 1607604
- [Background] Termanini B, Gibril F, Sutliff VE, Yu F, Venzon DJ, Jensen RT. Effect of long-term gastric acid suppressive therapy on serum vitamin B12 levels in patients with Zollinger-Ellison syndrome. Am J Med. 1998 May;104(5):422-30. doi: 10.1016/s0002-9343(98)00087-4. PMID 9626024
- [Derived] Vanclooster A, van Deursen C, Jaspers R, Cassiman D, Koek G. Proton Pump Inhibitors Decrease Phlebotomy Need in HFE Hemochromatosis: Double-Blind Randomized Placebo-Controlled Trial. Gastroenterology. 2017 Sep;153(3):678-680.e2. doi: 10.1053/j.gastro.2017.06.006. Epub 2017 Jun 15. PMID 28624580